CLINICAL TRIAL: NCT03098849
Title: Effectiveness of a Buteyko-based Breathing Technique on Psycho-physiological Parameters of Adults With Asthma - a Randomized, Controlled Study
Brief Title: Effectiveness of a Buteyko-based Breathing Technique for Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RBT_10
Record Dates: First submitted 2017-03-10; First posted 2017-04-04 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Buteyko-based breathing technique training
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko Training (Experimental): Breathing exercises according to the Buteyko Breathing Technique
  Interventions: Other: Buteyko Breathing Technique
- Control Group (No Intervention): Standard care as usual

INTERVENTIONS:
Other: Buteyko Breathing Technique — Patients are trained in various exercises aiming at breath reduction and breath control as introduced by Dr. K. Buteyko
  Arms: Buteyko Training

SUMMARY:
The purpose of this study is to investigate the effects of a Buteyko-based breathing technique on physiological and psychological parameters in adults with asthma

DETAILED DESCRIPTION:
The investigators explore the effects of a Buteyko-based breathing technique training using a treatment group vs. control group design and a repeated measures design with follow-up measurements 3 and 6 months after the intervention. The sample size calculation was made for an effect of d = .20 with repeated measures, a power of 1- β = .80 and α = .05. Additionally the investigators plan to take measurements (only once) from healthy volunteers matching them (age and gender) with the asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, regular intake of prescribed asthma medication according to the AWMF scheme level 1, native speaker of german

Exclusion Criteria:

* Participation in another study, comorbidities (heart diseases, cancer still under treatment, psychiatric diseases)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Change in Endtidal CO2 | Between baseline and 3 month follow up
  Capnometry
Change in Nijmegen-Score | Between baseline and 3 month follow up
  Questionnare assessing hyperventilation
Change in Buteyko CP | Between baseline and 3 month follow up
  Breath hold test

SECONDARY OUTCOMES:
Spirometry: FEV1 | Between baseline and 3 month follow up
  FEV1
Spirometry: FEV1 | Between baseline and 6 month follow up
  FEV1
Spirometry: FEV1/VCin | Between baseline and 3 month follow up
  FEV1/VCin
Spirometry: FEV1/VCin | Between baseline and 6 month follow up
  FEV1/VCin
Spirometry: PEF | Between baseline and 3 month follow up
  PEF
Spirometry: PEF | Between baseline and 6 month follow up
  PEF
(untitled outcome) | Between baseline and 3 month follow up
  Oral exhaled Nitric oxide
(untitled outcome) | Between baseline and 6 month follow up
  Oral exhaled Nitric oxide
Heart Rate Variability (SDNN) | Between baseline and 3 month follow up
  SDNN
Heart Rate Variability (SDNN) | Between baseline and 6 month follow up
  SDNN
Heart Rate Variability (RMSSD) | Between baseline and 3 month follow up
  RMSSD
Heart Rate Variability (RMSSD) | Between baseline and 6 month follow up
  RMSSD
Heart Rate Variability (LF/HF) | Between baseline and 3 month follow up
  LF/HF
Heart Rate Variability (LF/HF) | Between baseline and 6 month follow up
  LF/HF
Vascular stiffness | Between baseline and 3 month follow up
  Pulse Wave Velocity
Vascular stiffness | Between baseline and 6 month follow up
  Pulse Wave Velocity
Blood Pressure | Between baseline and 3 month follow up
  Systolic and Diastolic
Blood Pressure | Between baseline and 6 month follow up
  Systolic and Diastolic
Haemodynamics Stroke volume | Between baseline and 3 month follow up
  Stroke volume
Haemodynamics Stroke volume | Between baseline and 6 month follow up
  Stroke volume
Haemodynamics Cardiac output | Between baseline and 3 month follow up
  Cardiac output
Haemodynamics Cardiac output | Between baseline and 6 month follow up
  Cardiac output
Haemodynamics Total Vascular Resistance | Between baseline and 3 month follow up
  Total Vascular Resistance
Haemodynamics Total Vascular Resistance | Between baseline and 6 month follow up
  Total Vascular Resistance
Haemodynamics Cardiac index | Between baseline and 3 month follow up
  Cardiac index
Haemodynamics Cardiac index | Between baseline and 6 month follow up
  Cardiac index
Haemodynamics Perfusion | Between baseline and 3 month follow up
  Perfusion index
Haemodynamics Perfusion | Between baseline and 6 month follow up
  Perfusion index
Haemodynamics Plethvariability | Between baseline and 3 month follow up
  Plethvariability index (PVI)
Haemodynamics Plethvariability | Between baseline and 6 month follow up
  Plethvariability index (PVI)
Oxygen Saturation | Between baseline and 3 month follow up
  SpO2
Oxygen Saturation | Between baseline and 6 month follow up
  SpO2
ACQ | Between baseline and 3 month follow up
  Asthma Control Questionnaire, E. Juniper
ACQ | Between baseline and 6 month follow up
  Asthma Control Questionnaire, E. Juniper
AQLQ | Between baseline and 3 month follow up
  Asthma Quality of Life Questionnaire, E. Juniper
AQLQ | Between baseline and 6 month follow up
  Asthma Quality of Life Questionnaire, E. Juniper
ARCIM Questionnaire | Between baseline and 3 month follow up
  Questionnaire focusing on respiratory complaints like mucus, snoring, blocked nose.
ARCIM Questionnaire | Between baseline and 6 month follow up
  Questionnaire focusing on respiratory complaints like mucus, snoring, blocked nose.
STAI Questionnaire | Between baseline and 3 month follow up
  State and Trait Anxiety Inventory
STAI Questionnaire | Between baseline and 6 month follow up
  State and Trait Anxiety Inventory
ASF Questionnaire | Between baseline and 3 month follow up
  "Aachener Selbstwirksamkeitsfragebogen"
ASF Questionnaire | Between baseline and 6 month follow up
  "Aachener Selbstwirksamkeitsfragebogen"
Asthma medication | Between baseline and 3 month follow up
  Kind and dosage of asthma specific medication like steroids or betamimetics
Asthma medication | Between baseline and 6 month follow up
  Kind and dosage of asthma specific medication like steroids or betamimetics

CONTACTS AND LOCATIONS:
Locations (1):
- ARCIM Institute, Filderstadt, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Vagedes K, Kuderer S, Ehmann R, Kohl M, Wildhaber J, Jorres RA, Vagedes J. Effect of Buteyko breathing technique on clinical and functional parameters in adult patients with asthma: a randomized, controlled study. Eur J Med Res. 2024 Jan 11;29(1):42. doi: 10.1186/s40001-023-01634-1. PMID 38212823